CLINICAL TRIAL: NCT01064063
Title: Randomized Controlled Clinical Evaluation to Compare Vanguard Cruciate Retaining and AGC Total Condylar Knee Implants
Acronym: Vanguard
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: East Sussex Hospitals NHS Trust (Other); Biomet U.K. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMETEU.CR.LEU29; NCT01064063 (Registry Identifier: Clinicaltrials.gov)
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Traumatic Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Patients will be randomised into two arms, one receiving the AGC CR cement knee system (control group), and the other receiving Vanguard CR cement knee system (trial group).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AGC knee (Active Comparator): Patients were randomised to receive an AGC Cruciate Retaining cement knee. This is the control group in the study; the AGC is the gold standard of Biomets' knee products.
  Interventions: Device: AGC knee
- Vanguard CR (Experimental): Patients were randomised to receive a Vanguard Cruciate Retaining Knee from the Vanguard system which encompasses concepts used in the AGC family of knees. The Vanguard is specifically designed to give greater knees stability through use of more anatomic patello-femoral kinematics.
  Interventions: Device: Vanguard CR

INTERVENTIONS:
Device: Vanguard CR — The Vanguard CR is a metal and polyethylene total condylar knee system. The system contains three primary components: femoral, tibial, and bearing components, and a peripheral component: the patella button.
  Arms: Vanguard CR
Device: AGC knee — The AGC knee is a metal and polyethylene total condylar knee system offering complete component interchangeability.
  Arms: AGC knee

SUMMARY:
This evaluation is being conducted on the relative new knee system, the Vanguard Cruciate Retaining (CR) to evaluate clinical efficacy of the Vanguard CR components.

DETAILED DESCRIPTION:
This clinical trial was initially designed as a multi-centre, randomized controlled study, comparing the Vanguard CR with the AGC in routine use. The study now is a single centre study.

The Vanguard CR system has been specifically designed to give greater knee stability through the use of more anatomic patello-femoral kinematics.

ELIGIBILITY:
Inclusion Criteria:

* Pre-op knee score of <70
* Scheduled to undergo primary total knee replacement with any of the following indication:

  1. pain and disabled knee joint resulting from Osteoarthritis, Rheumatoid Arthritis, or Traumatic arthritis.
  2. One or more compartments involved.
* Need to obtain pain relief and improve function
* Ability and willingness to follow instructions, including control of weight and activity level, and to return for follow-up evaluations
* A good nutritional state of the patient
* Full skeletal maturity of the patient, patients who are at least 18 years of age.
* Patients of either sex
* Consent form read, understood, and signed by patient

Exclusion Criteria:

* Pre-op knee score greater than or equal to 70
* Infection
* Osteomyelitis
* Previous partial or total prosthetic knee replacement on the operative side
* Skeletal immaturity of the patient, patients who are less than 18 years of age.
* Sepsis
* Uncooperative patient or patient with neurological disorders who are incapable of following directions
* Osteomalacia
* Distant foci of infections
* Rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy, or neuromuscular disease in affected limb
* Incomplete or deficient soft tissue surrounding the knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-02-15 (Actual); Primary Completion 2013-12-15 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
American Knee Society Knee Score | 2 year
  Objective scoring system to rate the knee and patient's functional abilities before and after TKA

SECONDARY OUTCOMES:
Patient success | 2 year
  Defined as Knee Score greater than or equal to 80, No component revisions or removals, No pending component revisions or removals, Absence of osteolysis, No migration/subsidence of >3mm or >3 degrees
American Knee Society Score, Oxford Knee-12, SF-12 | 6w, 6m, 1y, 2y, 3y, 5y, 7y, 10y
  Objective scoring instruments to rate the knee and patient's functional abilities before and after TKA including scoring systems based on patient questionnaires
Radiographic evaluation | 6m,1y, 2y, 3y, 5y, 10y
  Assessment of patient x-rays
Adverse Events | any
  Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including an abnormal laboratory finding) in subjects, users or other persons, whether or not related to the investigational medical device.
Survivorship | 10 years
  Implant survivorship based on removal of a study device.
Noble & Weiss Knee Score, Kujala Score | 6w, 6m, 1y, 2y
  Scoring systems based on patient questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: A. Butler-Manual, FRCS, Principal Investigator — East Sussex Hospital NHS Trust - Conquest Hospital
Locations (1):
- East Sussex Hospital NHS Trust, Saint Leonards-on-Sea, East Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No
To be confirmed.